CLINICAL TRIAL: NCT05695638
Title: Proseq Cancer: A Prospective Study of Comprehensive Genomic Profiling in Patients With Incurable Cancer in Search for Targeted Treatment
Brief Title: Proseq Cancer: Genomic Profiling in Patients With Incurable Cancer in Search for Targeted Treatment
Status: Recruiting | Type: Observational
Sponsor: Morten Ladekarl (Other)
Responsible Party: Sponsor-Investigator, Morten Ladekarl, Professor, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Other Study IDs: N-20200018
Record Dates: First submitted 2023-01-10; First posted 2023-01-25 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Solid Tumor, Unspecified, Adult; Haematological Malignancy
Keywords: Precision medicine; Personalized medicine; Genomic profiling; Tissue agnostic
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — For molecular profiling the tumor DNA is subjected to somatic short variant detection using tumor/normal WES analysis, detection of copy number alterations, TMB and MSI status, and mutational signature analysis. Tumor RNA is used for the generation of an expression profile. Moreover, RNAseq enables detection of fusion transcripts. ctDNA is extracted from 10 ml blood samples or peritoneal fluid. Sequencing is performed on a NovaSeq 6000. Clinically relevant pathogenic variants are detected in a small set of genes. Germline variants in other genes are not analyzed, unless specifically requested and consented by the patient. Raw sequencing data are processed and stored under the regional IT-system. Sequencing data and supplementary metadata are submitted to the Danish National Genome Center.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Intention-to-treat cohort: All patients included

SUMMARY:
Proseq Cancer is a precision medicine program based on in-house whole exome sequencing (WES) and RNA sequencing. The approved protocol allows for biobanking, registration of clinical and laboratory data, and sharing of genomic data with the purpose of research, while fulfilling the Danish General Data Protection Regulation (GDPR) requirements. Patients are recruited from the North Denmark Region.

Treatment can be offered on site if a targeted drug of a nationally approved indication is suggested by the national tumor board (NTB). If not, the patient may be treated in an available clinical protocol. If no approved drug or relevant protocol is available or feasible, treatment with a targeted drug used outside a clinical protocol is pursued.

DETAILED DESCRIPTION:
Patients are recruited from the North Denmark Region. This is a precision medicine program based on in-house whole exome sequencing (WES) and RNA sequencing (RNAseq). All eligible patients are offered enrollment in an approved protocol, which allows for biobanking, registration of clinical and laboratory data, and sharing of genomic data with the purpose of research, while fulfilling the Danish GDPR requirements.

After informed consent clinical-pathological baseline data is registered by oncological investigators. Results of new pathological and molecular assessments are prospectively registered as well as decisions made at the National molecular Tumor Board (NTB).

New 1.2 mm core needle biopsies are taken from the most easily accessible, preferably progressing tumor lesion that has not been irradiated, usually guided by ultrasound. Biopsies from centrally located lung lesions or other sites with increased risk of complications, or procedures requiring general anesthesia are generally avoided. In each case, one biopsy is fixed in neutral-buffered formalin and allocated to histopathological assessment. Another, adjacent 1-2 biopsies are kept in RNAlater until processing for molecular analysis within 5 days. Patients with intracranial tumors are biopsied at time of diagnostic surgery or if surgery is otherwise required, and tissue is kept frozen at -80°C until the clinical course indicates that patients are eligible for the protocol. In parallel, a 10 ml EDTA blood sample is drawn for analysis of non-tumoral DNA. Unfixed or fresh frozen tissue material is preferred. However, in selected patients for whom a new biopsy is unobtainable and no fresh frozen tissue is available, DNA is extracted from the most recent FFPE archival sample of tumor tissue. Cell-free tumor-DNA (ctDNA) from peripheral blood samples is used in cases with insufficient tissue for analysis. Samples for ctDNA analysis are collected in cell-free DNA blood collection tubes (Streck).

The FFPE tumor biopsies are cut into four sections of 4 µm and one of 1 µm. One 4 µm section is stained with hematoxylin and eosin and another with HER2-antibody. The cancer and histological subtype are diagnosed by senior consultant pathologists. Additional pathological analyses, including immunohistochemistry or targeted NGS, are done on FFPE tissue at the initiative of the pathologist, or if requested by investigators or the tumor board.

The molecular profiling is performed in-house, but may also be performed at other sites. The in house procedure is as follows: Tissue biopsies in RNAlater or fresh frozen tissue are homogenized, and RNA and DNA is extracted using Qiagen AllPrep®. Non-tumoral DNA for profiling is extracted from peripheral blood leukocytes using QiaSymphony DSP DNA midi kit (Qiagen). WES library preparation is performed using the Sureselect XT HS Library Prep Kits (Agilent). Exome capture is performed using the SureSelect XT HS Clinical Research Exome V2 (Agilent), while RNAseq library preparation is done using the TruSeq Stranded mRNA Library Prep Kit (Illumina). Sequencing is carried out as 2x150 bp paired-end on a NovaSeq 6000 (Illumina), producing minimum 26 Gb, 18 Gb, or 33 million reads of raw sequence data for tumor DNA, non-tumoral DNA, or tumor RNA samples, respectively. For molecular profiling the tumor DNA is subjected to somatic short variant detection using tumor/normal WES analysis, detection of copy number alterations, TMB and MSI status, and mutational signature analysis. Tumor RNA is used for the generation of an expression profile used as input for tissue classification26. Moreover, RNAseq enables detection of fusion transcripts for identification of larger chromosomal abbreviations. ctDNA is extracted from 10 ml blood samples or, in few cases, from peritoneal fluid in cell-free DNA blood collection tubes (Streck) using QiaSymphony Virus/pathogen Midi Kit (Qiagen). TruSight Oncology 500 assay (Illumina) is used for library preparation. 2x150 bp paired-end sequencing is performed on a NovaSeq 6000 (Illumina) producing minimum 1500x coverage of the targeted regions.Using the non-tumoral DNA, clinically relevant pathogenic variants are detected in a small set of genes (BRCA1, BRCA2, ATM, MLH1, MSH2, MSH3, PMS1, MLH3, MSH6, PMS2, PALB2, RAD51C, RAD51D, MBD4, ANKRD26, CEBPA, DDX41, ETV6, GATA3, RUNX1, TERC, TERT and TP53). Germline variants in other genes are not analyzed, unless specifically requested by clinical geneticists and consented by the patient. Raw sequencing data are processed and stored under the regional IT-system. Sequencing data and supplementary metadata are submitted to the Danish National Genome Center. The in house bioinformatic procedure is as follows: Using Genome Analysis Tool Kit (GATK) the process largely follows the GATK-recommendations. The filtered variant file (VCF) is uploaded together with information on sex, age, diagnosis and detected fusion transcripts, gene losses or gains, to Qiagen Clinical Insight Interpret (QCI) for automatic classification of variants. All variants of clinical significance are manually verified by visual inspection of the DNA and RNAseq data. Variants are classified as pathogenic, likely pathogenic, variants of unknown significance (VUS), or benign/likely benign. QCI is also used prospectively to link variants and approved treatments or clinical trials into tiers. Non-tumoral variants are classified according to the 2015 ACMG/AMP guidelines and are, together with the history of patients, reviewed by an MD specialized in clinical genetics. If a germline variant with a likely consequence for the health of the patient or a relative is identified, patients who had requested this information at protocol consent are offered referral to the Department of Clinical Genetics. Reports are generated using a dedicated platform (PrOnco) from clinical data stored in REDCap and variants data. The platform enables a tumor board report to be generated on demand or made accessible through an interactive interface.

Cases are presented at a weekly web-based multidisciplinary NTB, directed by the phase I unit at Rigshospitalet, Copenhagen. Based on patients' history and characteristics, disclosed molecular variants, gene signatures or other tumor characteristics and available trials or drugs, matched treatments and early phase clinical trials are suggested.

Treatment can be offered on site if a targeted drug of a nationally approved indication is suggested by the NTB. If not, the patient may be treated in an available clinical protocol. This especially includes the ProTarget trial - a nation-wide, investigator-initiated basket trial of targeted treatment, studying the efficacy of approved drugs used "off label" in cohorts of patients with a similar target, similar drug and similar diagnosis (NCT04341181). If no approved drug or relevant protocol is available or feasible, treatment with a targeted drug used outside a clinical protocol is pursued. This includes treatment with a drug that is labelled but not approved by the Danish authorities, however, may be used after individual permission. It also includes "off label" treatment after individual permission, or "compassionate use" with an unapproved drug in a "named user program". Patients treated with matched targeted drugs outside a clinical drug trial are evaluated by CT- or MR-scans and biomarkers at baseline and every 8th or 9th week until progression. Blood samples for research are drawn and stored in Bio-and Genome Bank Denmark, while treatment data is registered prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Incurable, progressing and/or life-threatening cancer
* Expected residual survival of at least 3 months
* No efficient remaining standard treatment options
* Patient recruited from the Region of Northern Jutland, Denmark

Exclusion Criteria:

* WHO Performance Status >2
* Significant comorbidity, concurrent medication or laboratory values imposing an unacceptable risk at medical oncological treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with incurable, progressing and/or life-threatening cancer with an expected residual survival of at least 3 months and no efficient remaining standard treatment options. Patients are recruited from the Region of Northern Jutland, Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2030-05-31 (Estimated); Study Completion 2035-05-31 (Estimated)

PRIMARY OUTCOMES:
The fraction (in %) of patients having a tumor molecular profiling done, for whom a molecularly "druggable" variant can be identified | 10 years
  Total number of patients included for whom a molecular variant can be identified that potentially can be matched with a targeted drug, labelled for use in cancer, divided by total number of patients included having a tumor molecular profiling done.

CONTACTS AND LOCATIONS:
Overall Officials: Morten Ladekarl, MD, DMSCi, Principal Investigator — Department of Oncology, Aalborg University Hospital, Denmark
Locations (1):
- Department of Oncology, Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ladekarl M, Nohr AK, Sonderkaer M, Dahl SC, Sunde L, Vestereghem C, Mapendano CK, Haslund CA, Pagh A, Carus A, Lorincz T, Nowicka-Matus K, Poulsen LO, Laursen RJ, Dybkaer K, Poulsen BK, Frokjaer JB, Brugmann AH, Ernst A, Wanders A, Bogsted M, Pedersen IS. Feasibility and early clinical impact of precision medicine for late-stage cancer patients in a regional public academic hospital. Acta Oncol. 2023 Mar;62(3):261-271. doi: 10.1080/0284186X.2023.2185542. Epub 2023 Mar 11. PMID 36905645
- [Derived] Jakobsen MZ, Torp EA, Issa II, Hoholt H, Sonderkaer M, Madsen J, Christensen LM, Jorgensen MP, Nohr AK, Brondum RF, Kristensen DT, Dybkaer K, Severinsen MT, Due H. Evaluation of reference sample type for somatic variant calling in myeloid cancers. Ann Hematol. 2025 Nov;104(11):6091-6095. doi: 10.1007/s00277-025-06699-y. Epub 2025 Oct 22. PMID 41123648